CLINICAL TRIAL: NCT00401531
Title: Immunogenicity Study of a DTaP IPV Hep B PRP T Combined Vaccine in Comparison to Infanrix Hexa™, Both Concomitantly Administered With Prevnar™ at 2, 4, and 6 Months of Age in Thai Infants
Brief Title: Comparison of a DTaP-IPV-HB-PRP~T Combined Vaccine to Infanrix™-Hexa, When Administered With Prevnar® in Thai Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: A3L12
Record Dates: First submitted 2006-11-16; First posted 2006-11-20 (Estimated); Results first posted 2014-04-01 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-02

CONDITIONS: Hepatitis B; Polio; Diphtheria; Pertussis; Haemophilus Influenzae Type b
Keywords: Hepatitis B; Polio; Diphtheria; Pertussis; H. influenzae type b
MeSH Terms: conditions — Hepatitis B; Poliomyelitis; Diphtheria; Whooping Cough; Haemophilus Infections | interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: DTaP IPV Hep B PRP T + Prevnar™ (Experimental)
  Interventions: Biological: DTaP-IPV-HB-PRP~T and Pneumococcal polysaccharide vaccines
- Group 2: Infanrix hexa™ + Prevnar™ (Active Comparator)
  Interventions: Biological: DTaP-HB-IPV and Pneumococcal polysaccharide vaccines

INTERVENTIONS:
Biological: DTaP-IPV-HB-PRP~T and Pneumococcal polysaccharide vaccines — 0.5 mL, IM
  Other Names: Prevnar®
  Arms: Group 1: DTaP IPV Hep B PRP T + Prevnar™
Biological: DTaP-HB-IPV and Pneumococcal polysaccharide vaccines — 0.5 mL, IM
  Other Names: Infanrix™-Hexa; Prevnar®
  Arms: Group 2: Infanrix hexa™ + Prevnar™

SUMMARY:
The purpose of the study is to provide immunogenicity and safety data of the investigational hexavalent vaccine when it is given concomitantly (the same day at separate injection sites) with Prevnar, according to the 2-4-6 month immunization schedule, following one dose of HB vaccine at birth.

Primary Objective:

To demonstrate that the hexavalent DTaP-IPV-HB-PRP~T combined vaccine induces an immune response that is at least as good as the response following Infanrix™-Hexa in terms of seroprotection rates to HB and PRP, one month after a 3 dose primary series (2, 4, and 6 months), when co-administered with Prevnar®

Secondary Objectives:

Immunogenicity:

To describe in each group the immunogenicity parameters to each vaccine component (for DTaP-IPV-HB-PRP~T and Infanrix™-Hexa) one month after the third dose of the primary series.

Safety:

To describe the overall safety after each injection.

ELIGIBILITY:
Inclusion Criteria :

* Two month old infant (50 to 71 days old) on the day of inclusion, of either gender.
* Born at full term of pregnancy (>= 37 weeks) and with a birth weight >= 2.5 kg.
* Hepatitis B vaccination since birth.
* Informed consent form signed by one parent/legally acceptable representative and an independent witness if the parent/legally acceptable representative is illiterate.
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria :

* Participation in another clinical trial in the 4 weeks preceding the first trial vaccination.
* Planned participation in another clinical trial during the present trial period.
* Systemic hypersensitivity to any of the vaccine components or history of a life threatening reaction to the trial vaccine or a vaccine containing the same substances.
* Congenital or acquired immunodeficiency, or immunosuppressive therapy such as long-term systemic corticosteroid therapy.
* Chronic illness at a stage that could interfere with trial conduct or completion.
* Blood or blood-derived products received since birth.
* Any vaccination in the 4 weeks preceding the first trial vaccination.
* Any planned vaccination (except trial vaccinations) during the trial.
* Documented history of pertussis, T, D, polio, Hib, hepatitis B or Streptococcus pneumoniae infection(s) (confirmed either clinically, serologically, or microbiologically).
* Previous vaccination against pertussis, tetanus, diphtheria, poliomyelitis, Haemophilus influenzae type b infection(s) or Streptococcus pneumoniae.
* Known personal or maternal history of HIV, HB (HbsAg carrier) or hepatitis C seropositivity.
* Known thrombocytopenia or bleeding disorder contraindicating IM vaccination.
* History of seizures.
* Febrile (rectal equivalent temperature >= 38.0°C) or acute illness on the day of inclusion.

Ages: 50 Days to 71 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 412 (Actual)
Dates: Start 2006-10; Primary Completion 2007-11 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (2):
- Thailand (2):
  - Bangkok
  - Khonkaen

REFERENCES:
- [Result] Kosalaraksa P, Thisyakorn U, Benjaponpitak S, Chokephaibulkit K, Santos-Lima E. Immunogenicity and safety study of a new DTaP-IPV-Hep B-PRP-T combined vaccine compared to a licensed DTaP-IPV-Hep B//PRP-T comparator, both concomitantly administered with a 7-valent pneumococcal conjugate vaccine at 2, 4, and 6 months of age in Thai infants. Int J Infect Dis. 2011 Apr;15(4):e249-56. doi: 10.1016/j.ijid.2010.12.004. Epub 2011 Feb 18. PMID 21334243
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 22 October 2006 to 19 November 2007 in 4 clinical centers in Thailand.
Pre-assignment Details: A total of 412 participants who met all the inclusion, but none of the exclusion criteria were enrolled and vaccinated.
Groups:
- DTaP-IPV-Hep B-PRP-T + Prevnar™: Participants received a 3-dose primary vaccination series of diphtheria, tetanus, pertussis (2 component acellular), recombinant hepatitis B Hansenula and poliovirus vaccine adsorbed, and Haemophilus influenzae type B vaccine, conjugated to tetanus protein (DTaP-IPV-Hep B-PRP-T) vaccine co-administered with Prevnar vaccine (at 2, 4, and 6 months of age). All participants had received hepatitis B vaccination at birth.
- Infanrix Hexa™ + Prevnar™: Participants received a 3-dose primary vaccination series of Infanrix hexa vaccine co-administered with Prevnar vaccine (at 2, 4, and 6 months of age). All participants had received hepatitis B vaccination at birth.
Period: Overall Study
Arm/Group | DTaP-IPV-Hep B-PRP-T + Prevnar™ | Infanrix Hexa™ + Prevnar™
Started | 206 | 206
Completed | 197 | 196
Not Completed | 9 | 10
Not completed — Adverse Event | 2 | 0
Not completed — Protocol Violation | 3 | 7
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DTaP-IPV-Hep B-PRP-T + Prevnar™ | Infanrix Hexa™ + Prevnar™ | Total
Number analyzed (Participants) | 206 | 206 | 412
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 206 | 206 | 412
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months]
  Age Continuous | 1.88 (0.170) | 1.90 (0.187) | 1.89 (0.179)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 111 | 205
  Male | 112 | 95 | 207
Region of Enrollment [Number; unit: Participants]
  Thailand | 206 | 206 | 412

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Seroprotection Against Hepatitis B and Haemophilus Influenzae Type b Post-vaccination With Either DTaP-IPV-Hep B-PRP~T + Prevnar™ or Infanrix Hexa™ + Prevnar™
Description: Anti-Hepatitis B antibodies were measured using chemiluminescence detection technology; seroprotection was defined as a titer ≥ 10 mIU/mL. Anti-Haemophilus influenzae type b (anti-PRP) antibodies were measured by radioimmunoassay; seroprotection was defined as a titer ≥ 0.15 µg/mL.
Time Frame: Day 150 post-dose 1
Population: Seroprotection was assessed in the participants who had not committed any protocol violation that could have interfered with the primary criteria evaluation, per-protocol population.
Measure: Number; unit: Participants
Arm/Group | DTaP-IPV-Hep B-PRP-T + Prevnar™ | Infanrix Hexa™ + Prevnar™
Number analyzed (Participants) | 189 | 190
Participants
  Anti-Hepatitis B (N = 188, 190) | 187 | 189 [0 to 0]
  Anti-PRP (N = 189, 190) | 183 | 183 [0 to 0]

2. Secondary Outcome: Number of Participants With Seroprotection Against Diphtheria and Tetanus Post-vaccination With Either DTaP-IPV-Hep B-PRP~T + Prevnar™ or Infanrix Hexa™ + Prevnar™
Description: Anti-Diphtheria antibodies were measured by a toxin neutralization test. Anti-Tetanus antibodies were measured by an indirect enzyme-linked immunosorbent assay (ELISA). Seroprotection was defined for both as a titer ≥ 0.01 IU/mL.
Time Frame: Day 150 post-dose 1
Population: Seroprotection was assessed in the participants who had not committed any protocol violation that could have interfered with the primary criteria valuation, per-protocol population.
Measure: Number; unit: Participants
Arm/Group | DTaP-IPV-Hep B-PRP-T + Prevnar™ | Infanrix Hexa™ + Prevnar™
Number analyzed (Participants) | 189 | 190
Participants
  Anti-Diphtheria | 184 | 190 [0 to 0]
  Anti-Tetanus | 189 | 190 [0 to 0]

3. Secondary Outcome: Number of Participants With Seroprotection Against Poliovirus Types 1, 2, and 3 Post-vaccination With Either DTaP-IPV-Hep B-PRP~T + Prevnar™ or Infanrix Hexa™ + Prevnar™
Description: Anti poliovirus types 1, 2, and 3 antibodies were measured by neutralization assay. Seroprotection was defined as a titer ≥ 8 1/dil
Time Frame: Day 150 post-dose 1
Population: Seroprotection was assessed in participants who had not committed any protocol violation that could have interfered with the primary criteria evaluation, per-protocol population.
Measure: Number; unit: Participants
Arm/Group | DTaP-IPV-Hep B-PRP-T + Prevnar™ | Infanrix Hexa™ + Prevnar™
Number analyzed (Participants) | 187 | 186
Participants
  Anti Polio Type 1 | 187 | 186 [0 to 0]
  Anti Polio Type 2 | 187 | 186 [0 to 0]
  Anti Polio Type 3 | 187 | 185 [0 to 0]

4. Secondary Outcome: Number of Participants With Seroconversion Against Pertussis Post-vaccination With Either DTaP-IPV-Hep B-PRP~T + Prevnar™ or Infanrix Hexa™ + Prevnar™
Description: Anti pertussis toxoid (PT) and anti-filamentous hemagglutinin (FHA) antibodies were measured by enzyme linked immunosorbent assay (ELISA). Seroconversion was defined as ≥ 4 fold increase over baseline.
Time Frame: Day 150 post-dose 1
Population: Seroconversion was assessed in participants who had not committed any protocol violation that could have interfered with the primary criteria evaluation per-protocol population.
Measure: Number; unit: Participants
Arm/Group | DTaP-IPV-Hep B-PRP-T + Prevnar™ | Infanrix Hexa™ + Prevnar™
Number analyzed (Participants) | 189 | 190
Participants
  Anti-pertussis toxoid (N = 189, 189) | 177 | 177 [0 to 0]
  Anti-Filamentous hemagglutinin (N = 187, 188) | 177 | 179 [0 to 0]

5. Secondary Outcome: Geometric Mean Titers (GMTs) of Vaccine Antibodies Post-vaccination With Either DTaP-IPV-Hep B-PRP~T + Prevnar™ or Infanrix Hexa™ + Prevnar™
Description: Anti-hepatitis B antibodies were measured using chemiluminescence detection technology. Anti-Haemophilus influenzae type b (anti-PRP) antibodies were measured by radioimmunoassay, anti-Diphtheria by toxin neutralization assay, anti-Tetanus and anti-Pertussis by enzyme-linked immunosorbent assay (ELISA), and anti-Polio by neutralization assay.
Time Frame: Day 150 post-dose 1
Population: Antibody titers were assessed in participants who had not committed any protocol violation that could have interfered with the primary criteria evaluation, the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | DTaP-IPV-Hep B-PRP-T + Prevnar™ | Infanrix Hexa™ + Prevnar™
Number analyzed (Participants) | 189 | 190
Titers
  Anti-Hepatitis B (N = 188, 190) | 2477 [2044 to 3002] | 2442 [2096 to 2844]
  Anti-PRP (N = 189, 190) | 5.07 [4.05 to 6.33] | 2.41 [1.95 to 2.98]
  Anti-Diphtheria (N = 189, 190) | 0.297 [0.241 to 0.367] | 0.209 [0.177 to 0.247]
  Anti-Tetanus (N = 189, 190) | 1.38 [1.25 to 1.52] | 1.83 [1.69 to 1.97]
  Anti-Polio Type 1 (N = 187, 186) | 765 [649 to 902] | 1566 [1326 to 1850]
  Anti-Polio Type 2 (N = 187, 186) | 1489 [1259 to 1761] | 2277 [1905 to 2723]
  Anti-Polio Type 3 (N = 187, 186) | 837 [695 to 1007] | 2029 [1646 to 2502]
  Anti-Pertussis toxoid (N = 189, 189) | 168 [154 to 183] | 200 [185 to 216]
  Anti-Filamentous hemagglutinin (N = 188, 188) | 148 [136 to 162] | 123 [113 to 132]

6. Secondary Outcome: Number of Participants Reporting Solicited Injection Site and Systemic Reactions Post-vaccination With Either DTaP-IPV-Hep B-PRP~T + Prevnar™ or Infanrix Hexa™ + Prevnar™
Description: Solicited Injection Site Reactions: Pain, Erythema, and Swelling. Solicited Systemic Reactions: Pyrexia, Vomiting, Crying, Somnolence, Anorexia, and Irritability Grade 3: Pain, cries when injected limb is moved or the movement of the injected limb is reduced; Erythema and Swelling, ≥5 cm.
  Grade 3: Pyrexia, >39°C; Vomiting, ≥6 episodes per 24 hours or requiring parenteral hydration; Crying, >3 hours; Somnolence, Sleeping most of the time or difficult to wake up; Anorexia, Refuses ≥3 feeds/meals or refuses most feeds/meals; and Irritability, Inconsolable.
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Solicited reactions were assessed in all participants that were enrolled and vaccinated, intent-to-treat population.
Measure: Number; unit: Participants
Arm/Group | DTaP-IPV-Hep B-PRP-T + Prevnar™ | Infanrix Hexa™ + Prevnar™
Number analyzed (Participants) | 206 | 206
Participants
  Pain Post-dose 1 | 161 | 135 [0 to 0]
  Pain Post-dose 2 | 136 | 118 [0 to 0]
  Pain Post-dose 3 | 119 | 112 [0 to 0]
  Pain Post-any dose | 180 | 166
  Grade 3 Pain Post-any dose | 20 | 12
  Erythema Post-dose 1 | 79 | 64 [0 to 0]
  Erythema Post-dose 2 | 93 | 91 [0 to 0]
  Erythema Post-dose 3 | 86 | 79 [0 to 0]
  Erythema Post-any dose | 121 | 114
  Grade 3 Erythema Post-any dose | 3 | 2
  Swelling Post-dose 1 | 59 | 34 [0 to 0]
  Swelling Post-dose 2 | 52 | 44 [0 to 0]
  Swelling Post-dose 3 | 34 | 32 [0 to 0]
  Swelling Post-any dose | 85 | 65
  Grade 3 Swelling Post-any dose | 1 | 1
  Pyrexia Post-dose 1 | 109 | 68 [0 to 0]
  Pyrexia Post-dose 2 | 84 | 79 [0 to 0]
  Pyrexia Post-dose 3 | 81 | 81 [0 to 0]
  Pyrexia Post-any dose | 152 | 131
  Grade 3 Pyrexia Post-any dose | 6 | 7
  Vomiting Post Dose 1 | 47 | 56 [0 to 0]
  Vomiting Post-dose 2 | 28 | 32 [0 to 0]
  Vomiting Post-dose 3 | 22 | 28 [0 to 0]
  Vomiting Post-any dose | 77 | 82
  Grade 3 Vomiting Post-any dose | 1 | 3
  Crying Post-dose 1 | 128 | 106 [0 to 0]
  Crying Post-dose 2 | 106 | 104 [0 to 0]
  Crying Post-dose 3 | 77 | 75 [0 to 0]
  Crying Post-any dose | 167 | 153
  Grade 3 Crying Post-any dose | 7 | 5
  Somnolence Post-dose 1 | 109 | 104 [0 to 0]
  Somnolence Post-dose 2 | 91 | 79 [0 to 0]
  Somnolence Post-dose 3 | 55 | 59 [0 to 0]
  Somnolence Post-any dose | 141 | 125
  Grade 3 Somnolence post-any dose | 4 | 0
  Anorexia Post-dose 1 | 59 | 49 [0 to 0]
  Anorexia Post-dose 2 | 44 | 40 [0 to 0]
  Anorexia Post-dose 3 | 36 | 37 [0 to 0]
  Anorexia Post-any dose | 91 | 83
  Grade 3 Anorexia Post-any dose | 0 | 0
  Irritability Post-dose 1 | 134 | 122 [0 to 0]
  Irritability Post-dose 2 | 107 | 109 [0 to 0]
  Irritability Post-dose 3 | 90 | 88 [0 to 0]
  Irritability Post-any dose | 162 | 159
  Grade 3 Irritability Post-any dose | 4 | 6

ADVERSE EVENTS:
Time Frame: Adverse event data were collected following vaccination (Day 0) up to 10 months post-vaccination.
Arm/Group | DTaP-IPV-Hep B-PRP-T + Prevnar™ | Infanrix Hexa™ + Prevnar™
Serious Adverse Events (participants affected / at risk) | 6/206 | 8/206
Other Adverse Events (participants affected / at risk) | 161/206 | 135/206
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTaP-IPV-Hep B-PRP-T + Prevnar™ (N=206) | Infanrix Hexa™ + Prevnar™ (N=206)
Cryptorchism (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Eczema Herpeticum (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 3 (3)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Viral (Infections and infestations) | 1 (1) | 0 (0)
Urethritis (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Thermal Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Angioneurotic Oedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | DTaP-IPV-Hep B-PRP-T + Prevnar™ (N=206) | Infanrix Hexa™ + Prevnar™ (N=206)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 13 (13)
Vomiting (Gastrointestinal disorders) | 47/205 (47) | 56 (56)
Injection Site Pain (General disorders) | 161/205 (161) | 135 (135)
Injection Erythema (General disorders) | 93 (93) | 91 (91)
Injection Swelling (General disorders) | 59 (59) | 44 (44)
Irritability (General disorders) | 134/205 (134) | 122 (122)
Pyrexia (General disorders) | 109/205 (109) | 68 (68)
Nasopharyngitis (Infections and infestations) | 31 (31) | 35 (35)
Upper Respiratory Tract Infection (Infections and infestations) | 45 (45) | 46 (46)
Anorexia (Metabolism and nutrition disorders) | 59/205 (59) | 49 (49)
Somnolence (Nervous system disorders) | 109/205 (109) | 104 (104)
Crying (Psychiatric disorders) | 128 (128) | 106 (106)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications